CLINICAL TRIAL: NCT03255655
Title: Intense Therapeutic Ultrasound for Chronic Plantar Fascia Musculoskeletal Pain Reduction
Brief Title: Intense Therapeutic Ultrasound - Treatment for Chronic Plantar Fascia Musculoskeletal Pain Reduction
Acronym: ITU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guided Therapy Systems (Industry)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GTS - ITU UA Plantar Fascia 01
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Chronic Plantar Fasciitis
Keywords: Chronic Plantar Fasciitis; Plantar Fascia Pain; Intense Therapeutic Ultrasound (ITU); Guided Therapy Systems (GTS); Ardent Sound, Inc.; Actisound
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: Adult Patients (age 18 - 85) of either gender diagnosed with chronic plantar fasciitis pain (>90 days) where Standard of Care treatments had failed to reduce pain.
Who Masked: Investigator
Masking Description: Investigator was blinded to the treated vs. control/sham treated patient identity and to the treated foot.
  Researchers were blinded to the Investigators physical exam finding and patient outcome measure reports
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- ITU Treatment (Experimental): Intense Therapeutic Ultrasound (ITU) treatment applied along the length and width of the Plantar Fascia: 350 - 5 Joule pulses were applied twice, two weeks apart.
  Interventions: Device: Intense Therapeutic Ultrasound Treatment - ITU
- Sham ITU Treatment (Placebo Comparator): Sham / Placebo Intense Therapeutic Ultrasound treatment (ITU) applied along the length and width of the Plantar Fascia: 350 - 0 Joule pulses were applied twice, two weeks apart.
  Interventions: Device: Intense Therapeutic Ultrasound Treatment - ITU

INTERVENTIONS:
Device: Intense Therapeutic Ultrasound Treatment - ITU
  Other Names: Guided Therapy Systems, Ardent Sound, GTS, ITU

SUMMARY:
Double-blinded feasibility study for the treatment of pain related to chronic plantar fasciitis. A total 37 patients (27 treated and 12 control/sham treated) received 2 treatments, 2 weeks apart on subcutaneous plantar fascia musculoskeletal tissue along with Standard of Care treatments as prescribed by the Principal Investigator. Patients were followed for up to 6 months after the first treatment receiving a physical exam at each follow-up visit (4, 8 and 12 weeks) and provided feedback via Patient/Subject Reported Outcome Measure surveys specific to the treated anatomy at each visit and via phone follow-up at 26 weeks after the first treatment.

DETAILED DESCRIPTION:
Intense therapeutic ultrasound (ITU) is an established ultrasound based therapy in which sound waves are concentrated and focused into selected musculoskeletal tissue, to produce selective thermal coagulative changes over a small controlled area while leaving the surrounding tissue unaffected. These coagulative changes are known to begin the body's tissue response cascade and promote collagen generation in the targeted anatomy resulting in pain reduction.

ITU has been used clinically for treating the subcutaneous musculoskeletal tissue below facial skin for the past decade and it has received CE Mark and FDA 510(k) clearance to market for non-surgical brow and submental tissue lifting. Over 3 Million patients worldwide have been treated using this technology. Clinical studies have shown that 85% of patients receiving this treatment on facial skin tissue showed an improvement in facial lifting with no significant pain, erythema, inflammation or scarring by creating the same coagulative changes to the connective tissue under the skin. Histologically, it has been shown that ITU induces the production of dermal collagen with thickening of the dermis and straightening of the elastic fibers in the reticular dermis.

On-going research in laboratory studies has shown that ITU can improve healing of damaged Achilles tendon in a rabbit model. Preliminary results showed an increase in precursor markers for collagen regeneration (e.g. Vascular endothelial growth factor A (VEGFa), tumor necrosis factor alpha (TNFα), Interleukin 1 beta (IL-1β), and Transforming growth factor beta 1 (TGFβ1)) and subsequent increase in collagen formation in injured rabbit tendons treated with ITU compared to injured, untreated rabbit tendons.

ELIGIBILITY:
Inclusion Criteria:

* • Chronic Pain (>90 days) from previously diagnosed Plantar Fasciitis, where "Standard of Care" regimens failed to relief pain in the affected anatomy.

  * No History of surgery to the affected anatomy.
  * No alternative treatment procedures within the last 90 days.
  * Unilateral Pain
  * Willingness to complete treatment and post treatment regimen as described.
  * Patients who have provided written and verbal informed consent

Exclusion Criteria:

* • Patients currently enrolled in any other non-conservative, device, or Investigational New Drug clinical trial, or who have participated in a clinical study involving the Plantar Fascia, thirty days prior to study initiation;

  * Patients who have participated in any other clinical study involving an investigational product 30 days prior to enrollment that, in the opinion of the Principal Investigator, could affect the outcome of this study;
  * Patients who have received previous treatment in the symptomatic limb (not including conservative treatment);
  * At the Principal Investigator's discretion, any patient that should be excluded based on their current condition or medical history.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Latt, Md, Ph.D., Principal Investigator — University of Arizona; Orthopaedic Surgery and Biomedical Engineering; Department of Orthopaedic Surgery
Locations (1):
- The Univesity of Arizona; Orthopaedic Surgery and Biomedical Engineering, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White WM, Makin IR, Barthe PG, Slayton MH, Gliklich RE. Selective creation of thermal injury zones in the superficial musculoaponeurotic system using intense ultrasound therapy: a new target for noninvasive facial rejuvenation. Arch Facial Plast Surg. 2007 Jan-Feb;9(1):22-9. doi: 10.1001/archfaci.9.1.22. PMID 17224484
- [Background] Alam M, White LE, Martin N, Witherspoon J, Yoo S, West DP. Ultrasound tightening of facial and neck skin: a rater-blinded prospective cohort study. J Am Acad Dermatol. 2010 Feb;62(2):262-9. doi: 10.1016/j.jaad.2009.06.039. PMID 20115948
- [Background] Gliklich RE, White WM, Slayton MH, Barthe PG, Makin IR. Clinical pilot study of intense ultrasound therapy to deep dermal facial skin and subcutaneous tissues. Arch Facial Plast Surg. 2007 Mar-Apr;9(2):88-95. doi: 10.1001/archfaci.9.2.88. PMID 17372061
- [Background] Laubach HJ, Makin IR, Barthe PG, Slayton MH, Manstein D. Intense focused ultrasound: evaluation of a new treatment modality for precise microcoagulation within the skin. Dermatol Surg. 2008 May;34(5):727-34. doi: 10.1111/j.1524-4725.2008.34196.x. PMID 18429926
- [Background] Molloy T, Wang Y, Murrell G. The roles of growth factors in tendon and ligament healing. Sports Med. 2003;33(5):381-94. doi: 10.2165/00007256-200333050-00004. PMID 12696985
- [Background] DiGiovanni BF, Nawoczenski DA, Lintal ME, Moore EA, Murray JC, Wilding GE, Baumhauer JF. Tissue-specific plantar fascia-stretching exercise enhances outcomes in patients with chronic heel pain. A prospective, randomized study. J Bone Joint Surg Am. 2003 Jul;85(7):1270-7. doi: 10.2106/00004623-200307000-00013. PMID 12851352

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients 18 - 85 years previously diagnosed with unilateral Chronic Plantar Fasciitis (>90 days), where Standard of Care therapies had failed to reduce pain.
Groups:
- ITU Treatment for Chronic Plantar Fasciitis: Intense Therapeutic Ultrasound (ITU) treatment applied along the length and width of the Plantar Fascia: 350 - 5 Joule pulses were applied twice, two weeks apart.
  Intense Therapeutic Ultrasound Treatment - ITU
- Sham ITU Treatment for Chronic Plantar Fasciitis: Sham / Placebo Intense Therapeutic Ultrasound treatment (ITU) applied along the length and width of the Plantar Fascia: 350 - 0 Joule pulses were applied twice, two weeks apart.
  Intense Therapeutic Ultrasound Treatment - ITU
Period: Overall Study
Arm/Group | ITU Treatment for Chronic Plantar Fasciitis | Sham ITU Treatment for Chronic Plantar Fasciitis
Started | 29 | 12
Completed | 22 | 8
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ITU Treatment for Chronic Plantar Fasciitis | Sham ITU Treatment for Chronic Plantar Fasciitis | Total
Number analyzed (Participants) | 29 | 12 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 11 | 39
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 54 [35 to 83] | 47 [34 to 83] | 51 [34 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 8 | 32
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29 | 12 | 41

OUTCOME MEASURES:

1. Primary Outcome: Average Percentage of Change as Reported Using Foot Function Index Pain Subscale
Description: Average Percentage of Change as Reported using Foot Function Index (FFI) pain subscale. Range (±100%). Foot Function Index pain subscale is a measure of pain and disability and activity limitation based 9 questions, each with a possible pain score of 0 - 10, where 0 indicates no pain during the described activity and 10 indicates the worst imaginable pain during a described activity. A summed total score of 0 indicates the patient had no pain for all activities. A score of 90 indicates the patient experiences the worst imaginable pain for all the described activities. The results compare the average percentage change of the FFI score at 12 weeks, compared to the average FFI score at baseline.
Time Frame: 12 weeks after 1st Treatment
Population: Total population of respondents at 12 weeks.
Measure: Mean (Full Range); unit: percentage of Change
Arm/Group | ITU Treatment for Chronic Plantar Fasciitis | Sham ITU Treatment for Chronic Plantar Fasciitis
Number analyzed (Participants) | 22 | 8
percentage of Change | -54 [-100 to 100] | -25 [-100 to 100]

2. Primary Outcome: Mean Percentage Change in Volume of Plantar Fascia Hypoechoic Lesions by Diagnostic Ultrasound Imaging
Description: Mean Percentage Change in Volume of Plantar Fascia Hypoechoic Lesions by Diagnostic Ultrasound Imaging compared to Baseline Volume, where volume is calculated using: (4/3)π x R1 x R2 x R3, where R = Radius of each measurement: Lesion Length (1), Width (2), Depth (3).
Time Frame: 12 Weeks after the first Treatment
Population: Male and Female previously diagnosed with Chronic Plantar Fasciitis, between the age of 18 and 85.
Measure: Mean (Standard Error); unit: percentage of Hypoechoic Lesion Change
Arm/Group | ITU Treatment for Chronic Plantar Fasciitis | Sham ITU Treatment for Chronic Plantar Fasciitis
Number analyzed (Participants) | 22 | 8
percentage of Hypoechoic Lesion Change | -81 (8) | 26 (4)

ADVERSE EVENTS:
Time Frame: 2 years, 9 months
Description: Any Patient Self-Reported Adverse Event occurring during the treatment or during the Follow-up Period.
Arm/Group | ITU Treatment for Chronic Plantar Fasciitis | Sham ITU Treatment for Chronic Plantar Fasciitis
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/12
Other Adverse Events (participants affected / at risk) | 0/29 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2014-04-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT03255655/Prot_000.pdf
  • Informed Consent Form (2014-05-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT03255655/ICF_001.pdf
  • Statistical Analysis Plan (2014-05-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT03255655/SAP_002.pdf